CLINICAL TRIAL: NCT05710094
Title: Single-centre, Randomised, Double-blinded, Placebo-controlled Ascending Single Doses of SoftOx Biofilm Eradicator (SBE) and Open-label Once-, Twice-, and Thrice-daily Dosing of SBE for Five Days in Patients With Chronic Leg Wounds.
Brief Title: Safety and Tolerability of Single and Multiple Doses of SoftOx Biofilm Eradicator (SBE) in Chronic Leg Wounds
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SoftOx Solutions AS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SBE-01
Record Dates: First submitted 2021-10-18; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Chronic Leg Ulcer; Venous Leg Ulcer
Keywords: lower extremities infection biofilm antimicrobial
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Intervention Model Description: Randomised, double-blinded, placebo-controlled ascending single dose groups (Groups 1 to 4); followed by open-label multiple ascending dose groups (Groups 5 to 7)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinding and unblinding procedures applied only to the single-dose groups, i.e., Groups 1-4, randomized to receive SBE (active) or sterile saline (placebo).
  The computer-generated randomisation list was kept strictly confidential, accessible only to authorised persons, until the time of unblinding of the study.
  The following procedures were implemented in the single-dose groups to minimise the risk of unintended unblinding:
  i. Blinded staff prepared the patient's leg wound for the administration of IMP.
  ii. Both patient and blinded staff applied a nose clip, prior to and during IMP administration, until all materials used for the treatment (plastic wrapping, gauze, gallipot, etc.) had been removed and the room had been vented for a couple of minutes by opening a window.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Group 1 (Experimental): Single dose of 500ppm HOCl + 1 % HAc, or placebo
  Interventions: Drug: SoftOx Biofilm Eradicator (Groups 1 to 7); Device: Sterile isotonic saline (Groups 1 to 4)
- Group 2 (Experimental): Single dose of 500ppm HOCl + 2 % HAc, or placebo
  Interventions: Drug: SoftOx Biofilm Eradicator (Groups 1 to 7); Device: Sterile isotonic saline (Groups 1 to 4)
- Group 3 (Experimental): Single dose of 500ppm HOCl + 3 % HAc, or placebo
  Interventions: Drug: SoftOx Biofilm Eradicator (Groups 1 to 7); Device: Sterile isotonic saline (Groups 1 to 4)
- Group 4 (Experimental): Single dose of 1000ppm HOCl + 3 % HAc, or placebo
  Interventions: Drug: SoftOx Biofilm Eradicator (Groups 1 to 7); Device: Sterile isotonic saline (Groups 1 to 4)
- Group 5 (Experimental): Multiple doses (OD for 5 days) of xppm HOCl + x% HAc#
  Interventions: Drug: SoftOx Biofilm Eradicator (Groups 1 to 7)
- Group 6 (Experimental): Multiple doses (BID for 5 days) of xppm HOCl + x% HAc#
  Interventions: Drug: SoftOx Biofilm Eradicator (Groups 1 to 7)
- Group 7 (Experimental): Multiple doses (TID for 5 days) of xppm HOCl + x% HAc#
  Interventions: Drug: SoftOx Biofilm Eradicator (Groups 1 to 7)

INTERVENTIONS:
Drug: SoftOx Biofilm Eradicator (Groups 1 to 7) — SBE is a water-based formulation containing hypochlorous acid (HOCl) at concentrations of 500-1000 µg/mL and acetic acid (HAc) at concentrations of 1-3 %. Both active ingredients are naturally occurring molecules and have a long history of safe use in medicinal products and in solutions approved as medical devices. Both molecules, exhibit broad-spectrum antimicrobial activity at the concentrations present in SBE. The antimicrobial effect of HOCl is rapid and powerful by acting on and disrupting the function of key microbial molecules such as proteins, lipids, and nucleic acids, while remaining safe to mammalian cells and not promoting the emergence of new resistant microbes. Moreover, HOCl is active against biofilms, and some studies suggest that HOCl may also increase oxygenation of the wound site leading to improved healing.
  Other Names: SS0350
Device: Sterile isotonic saline (Groups 1 to 4) — Sterile isotonic saline was used as placebo because it is part of standard of care, used as an irrigation solution at dressing change and has the same appearance as SBE
  Other Names: Irriflex
  Arms: Group 1; Group 2; Group 3; Group 4

SUMMARY:
Single-centre clinical study investigating the safety and tolerability of randomised, double-blinded, placebo-controlled ascending single doses of topically applied SoftOx Biofilm Eradicator (SBE) in patients with chronic leg wounds and of open-label once daily, twice daily, and thrice daily dosing of topically applied SBE for five days in patients with chronic leg wounds. The primary objective of the study is to assess the safety and tolerability of single and multiple doses of topically applied SBE in patients with chronic leg wounds. A secondary objective of the study is to assess changes in bacterial burden in the leg wound after treatment with SBE.

DETAILED DESCRIPTION:
The study enrolled subjects with chronic leg wounds, i.e., the intended target population for SBE.

The first part of the study aimed to identify the highest tolerated dose of SBE in a randomised, double-blind, and placebo-controlled manner with sequential evaluation of 4 single ascending doses. As a precaution, sentinel and staggered dosing was applied in the single-dose groups: the safety of two subjects treated on two different days (at least one of whom was treated with SBE) was reviewed before commencing dosing of the remaining subjects in a single-dose group (sentinel dosing), with an interval of at least 1 hour between the dosing of different subjects (staggered dosing). The starting dose of 500 µg/mL HOCl + 1% HAc was based on previous knowledge concerning the MIC and MBC of SBE and the results obtained in a 28-day, repeated-dose toxicology study in minipigs. The latter indicated that up to 1000 µg/mL + 3% HAc (the highest dose tested) was well-tolerated. Choosing 500 µg/mL HOCl + 1% HAc as the starting dose in the current study provided a safety factor of 2 for HOCl and a safety factor of 3 for HAc. The highest well-tolerated dose of SBE in the non-clinical toxicology study was chosen as the highest single dose to be evaluated in the current study. Dose-escalation steps in the single-dose groups were conservatively defined with escalation factors ranging from 1 to 2. Prior to dose escalation, blinded results were evaluated by the Safety Monitoring Committee (SMC).

The second part of the study aimed to evaluate the safety and tolerability of multiple dosing of SBE. The multiple-dose groups tested different dosing regimens with formulations determined by the SMC based on the safety and tolerability of the formulations evaluated in the first part of the study. Three multiple-dose groups (once-, twice-, and thrice-daily administrations) were planned.

ELIGIBILITY:
INCLUSION CRITERIA

To be eligible for this study, patients must fulfil all of the following criteria:

1. Male and female patients aged 18 and above at time of informed consent.
2. Chronic (present for at least 4 weeks) leg wound, as judged by the Investigator, with a size of at least 1 cm2 and maximally 100 cm2 (measured as the width x length) on the day of the (first) administration of IMP.
3. Patients must have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the study, including possible risks and adverse effects.

EXCLUSION CRITERIA

Patients are not eligible for this study if they fulfil any of the following exclusion criteria:

1. Any surgical or medical condition, including findings in the medical history or in the pre-study assessments, or any other significant disease, that in the opinion of the Investigator, constitutes a risk or a contraindication for the participation of the patient in the study or that could interfere with the study objectives, conduct, or evaluation at screening or time of the (first) administration of IMP.
2. Known or clinical suspicion of cancer in the leg wound at screening or time of the (first) administration of IMP, e.g., basal cell carcinoma or squamous cell carcinoma.
3. Clinical symptoms of COVID-19 or positive test for SARS-CoV-2 (testing according to local procedures) at screening or on the day of the (first) administration of IMP.
4. Clinical infection requiring systemic antibiotics at time of the (first) administration of IMP.
5. Severe ischaemia in the target leg at screening or time of the (first) administration of IMP defined as an ankle brachial index (ABI) < 0.5.
6. Necrotic tissue in leg wound at time of the (first) administration of IMP.
7. Clinically significantly reduced perception of sensation or pain assessed in proximity of the wound at screening.
8. A pain score from the leg wound above 4 assessed on a 10 cm VAS , where 0 cm indicates no pain at all and 10 cm indicates the worst imaginable pain at time of the (first) administration of IMP.
9. Use of opioids from time of screening to end of study, unless used a at stable dose, as judged by the Investigator.
10. Participation in the treatment phase of a clinical study with an investigational new drug within 30 days or 5 half-lives (whichever is longer) before the (first) administration of IMP.
11. Has previously received SBE in any of the concentrations tested in the current study.
12. Pregnant or lactating at screening or time of the (first) administration of IMP.
13. Ascertained or presumptive allergy/ hypersensitivity to any components of the IMP; history of anaphylaxis to drugs or serious allergic reactions leading to hospitalisation or any other allergy reaction in general, which the Investigator considers may affect the safety of the patient and/or outcome of the study.
14. Inability to communicate or cooperate with the Investigator (e.g., language problems, illiteracy, poor mental status) or to comply with the requirements of the study.
15. Other factors which in the opinion of the Investigator may interfere with study conduct.
16. Legal incapacity or limited legal capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Nature, occurrence, and severity of adverse events (AEs) | From the start of the first administration of IMP to 3 to 5 days after the last administration of IMP
  Clinically significant abnormal values of vital signs (systolic and diastolic blood pressure, pulse rate, respiratory rate, body temperature), safety blood and urine parameters, ECG, and physical examination will be reported as AEs.
Change from baseline in wound pain assessed by use of visual analogue scale (VAS). | From the start of the first administration of IMP to 3 to 5 days after the last administration of IMP
  Change from baseline i.e., the last value before the (first) administration of IMP, in wound pain as assessed by use of a 10 cm VAS, where 0 cm indicated no pain at all, and 10 cm indicated the worst imaginable pain at the time of assessment.

SECONDARY OUTCOMES:
Change from baseline in wound bacterial burden (number of colony-forming units per mL; CFU/mL) | From the start of the first administration of IMP to 3 to 5 days after the last administration of IMP
  The bacterial burden of wounds was assessed using surface swabs (collected with the Z technique) at baseline, i.e., before the first administration of IMP, 20 min after the administration of IMP (on the treatment day for the single-dose groups, on each day of treatment for the OD multiple-dose group and after the second administration on each day of treatment for the BID multiple-dose group) and at the Follow-up visit.

OTHER OUTCOMES:
Change from baseline in wound area | From the start of the first administration of IMP to 3 to 5 days after the last administration of IMP
  The area of the wound in cm2 was calculated by the width x length (both in cm) of the wound. Wound area was estimated at screening, at baseline, i.e., before the (first) administration of IMP, and at the Follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: David Peick Sonne, MD; PhD, Principal Investigator — Bispebjerg and Frederiksberg Hospital; Glenn Gundersen, PhD, Study Director — SoftOx Solutions A/S
Locations (1):
- Bispebjerg University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No